CLINICAL TRIAL: NCT05141630
Title: Safety of Axillary Sentinel or Targeted Lymph Node Biopsy Alone After Neoadjuvant Chemotherapy in Breast Cancer With Initial Axillary Metastasis
Brief Title: Axillary Sentinel or Targeted Lymph Node Biopsy Alone After Neoadjuvant Chemotherapy in Node-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Department of Breast Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTLEY
Record Dates: First submitted 2021-11-08; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; neoadjuvant chemotherapy; axillary nodal management
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group with axillary sentinel or targeted lymph node biopsy alone (Experimental): The patients with stage II to III breast cancer with biopsy-confirmed nodal metastases who convert to cN0 following NAC is recruited. Eligible patients are treated with axillary sentinel or targeted lymph node biopsy alone. Post-surgery radiation therapy will be administered at the discretion of the radiologist and the nodal radiotherapy must be conducted in patients with low nodal disease.
  Interventions: Procedure: sentinel lymph node biopsy or targeted axillary dissection alone

INTERVENTIONS:
Procedure: sentinel lymph node biopsy or targeted axillary dissection alone — sentinel lymph node biopsy or targeted axillary dissection alone

SUMMARY:
This randomized phase II trial investigates the effectiveness of axillary sentinel or targeted lymph node biopsy alone after neoadjuvant chemotherapy (NAC) in breast cancer patients with initial axillary metastasis. For patients with the low nodal disease after NAC, it is not yet known if radiation therapy causes fewer side effects without compromising loco-regional control.

DETAILED DESCRIPTION:
To evaluate long-term survival and life quality in patients with biopsy-proven node-positive (cN1-N2) breast cancer receiving NAC, followed by limited nodal burden (less than two positive lymph nodes) by using a (sentinel lymph node biopsy) SLNB or targeted axillary dissection (TAD) technique, and no further axillary surgery.

OUTLINE:

Eligible patients with cT1 to cT3 biopsy-proven N1-2 breast cancer rendered cN0 by NAC underwent SLNB with dual tracer mapping or TAD, and omission of ALND if 2 or more biopsied nodes were identified and less than 2 biopsied nodes were pathologically positve. Metastatic nodes were not routinely clipped, and localization of clipped nodes was performed in these patients. The study was performed in a single cancer center.

After study treatment, patients are followed up at least every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study within 10 years.

ELIGIBILITY:
Pre-Registration Eligibility Criteria:

1. Clinical stage T1-3 N1-2M0 breast cancer at diagnosis (prior to neoadjuvant chemotherapy) by American Joint Committee on Cancer (AJCC) staging 7th edition 2. No inflammatory breast cancer 3. No other malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix 4. All patients must have had an axillary ultrasound with fine needle aspiration (FNA) or core needle biopsy (CNB) of axillary lymph nodes documenting axillary metastasis at the time of diagnosis, prior to or at most 14 days after starting neoadjuvant chemotherapy (NAC)

* Note: Biopsy of intramammary nodes does not fulfill eligibility criteria; In some patients, a clip is implanted into positive lymph nodes verified by FNA or CNB under the guidance of ultrasound 5. Patients must have had estrogen receptor, progesterone receptor and HER2 status (by immunohistochemistry [IHC] and/or in situ hybridization [ISH]) evaluated on CNB prior to start of NAC
* Note: If HER2 status has not been clearly determined (i.e. equivocal/indeterminate), then patients should not be enrolled 6. Patients must have completed all planned cycles and regimens of NAC prior to surgery; sandwich chemotherapy is not allowed (i.e. anthracycline/cytoxan or taxane chemotherapy planned to be given after surgery); patients must have completed at least 4 cycles of NAC consisting of an anthracycline and/or taxane-based regimen without evidence of disease progression in the breast or the lymph nodes
* Note: Delays/dose modifications due to toxicities/adverse events are allowed as long as a minimum of 4 cycles of NAC is administered; more than 4 cycles of NAC may be administered at the discretion of the treating medical oncologist 7. Patients with HER-2 positive tumors must have received neoadjuvant trastuzumab, or trastuzumab + pertuzumab, or other approved anti-HER-2 therapy (either with all or with a portion of the NAC regimen); therapy must be Food and Drug Administration (FDA)-approved targeted anti-HER2 therapy, but additional therapies are allowed as are non-trastuzumab regimens if administered in the context of an Institutional Review Board (IRB)-approved clinical trial 8. All patients must have a clinically negative axilla (no bulky adenopathy) on physical examination documented at the completion of NAC
* Note: an ultrasound of the axilla is not required at completion of NAC; if performed, its findings do NOT impact eligibility 9. No more than 8 weeks of neoadjuvant endocrine therapy prior to the start of NAC 10. No neoadjuvant radiation therapy 11. No SLN surgery/excisional biopsy for pathological confirmation of axillary status prior to or during NAC 12. No prior history of ipsilateral breast cancer (invasive disease or ductal carcinoma in situ [DCIS]); lobular carcinoma in situ (LCIS) and benign breast disease is allowed 13. No prior ipsilateral axillary surgery, such as excisional biopsy of lymph node(s) or treatment of hidradenitis 14. No history of prior or concurrent contralateral invasive breast cancer; benign breast disease; LCIS or DCIS of contralateral breast is allowed 15. Patients must not be pregnant or nursing
* Note: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential 16. Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1

Intra-Operative Registration/Randomization Criteria:

1. Breast surgery (lumpectomy or mastectomy) and SLN or targeted axillary dissection (TAD) surgery must be completed within 30 days of the completion of the last dose of NAC
2. SLNB is rountinely performed after NAC using dual tracer mapping with technetium-99m sulfur colloid and isosulfan blue dye. Radioactive, blue, or palpably abnormal nodes were considered SLNs. In patients presenting with clips, localization of the clipped node was performed and surgeons were aware if the clipped node was retrieved during the SLNB.
3. A minimum of 2 and a maximum of 8 total nodes (sentinel + non-sentinel+/-clipped nodes) are identified and excised; more than 8 biopsied nodes identified by either surgeon or pathologist is not allowed Note: Patients who do not have an identifiable SLN will not be enrolled
4. Zero or one lymph node (sentinel + non-sentinel+/-clipped nodes) excised during SLNB or TAD with a metastasis identified on intra-operative pathologic assessment Note: Nodal macro/micro-metastasis (greater than 0.2 mm in greatest dimension) and isolated tumor cells (metastases less than or equal to 0.2 mm) will be treated as node positive disease (N0i+) Note: If on final pathology, more than 8 lymph nodes are seen pathologically, or two or more than two nodes turn positive pathologically, then the patient should not be recruited into the study.
5. Axillary lymph node dissection (ALND) is not to be performed prior to registration/randomization

Post-Operative Registration/Randomization Criteria:

1. For cases where ALND has not been performed and one of the following is true: 1) intra-operative evaluation of biopsied lymph node (including sentinel or non-sentinel or targeted nodes) turned to be negative and final pathology identified less than two positive lymph nodes with metastasis OR 2) biopsied lymph node considered negative on intra-operative evaluation was found to be positive on final pathology (only one positive lymph node is allowed)
2. Breast surgery (lumpectomy or mastectomy) and sentinel lymph node surgery must be completed within 30 days of the completion of the last dose of NAC; negative margin (by either breast conservation or mastectomy) on final pathology where negative margin is defined as no tumor on ink
3. For those patients who also undergo contralateral breast surgery, if invasive disease is found in the contralateral breast, the patient is not eligible for registration /randomization

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Nodal recurrence rate | Up to 5 years after completion of surgery (radiation therapy if done)
  a recurrence in the ipsilateral axillary, supraclavicular, or internalmammary nodal basins.

SECONDARY OUTCOMES:
Shoulder function as assessed by arm function test questionnaire at baseline, 1, 3, and 5 years after surgery | Up to 5 years after completion of surgery (radiation therapy if done)
Rate of patients who develop arm lymphedema if there is a 10% increase in the volume of the ipsilateral arm from its pre-surgery volume | Up to 5 years after completion of surgery (radiation therapy if done)
Invasive breast cancer recurrence-free interval | Up to 5 years after completion of surgery (radiation therapy if done)
  as the time from completion of radiation therapy until the date of first occurrence of one of the following events: ipsilateral invasive breast tumor, locoregional invasive disease, distant recurrence, contralateral invasive breast cancer, second primary invasive cancer.
Overall survival | Up to 5 years after completion of surgery (radiation therapy if done)
  as the time from completion of radiation therapy until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu SY, Li JW, Wang YJ, Jin KR, Yang BL, Li JJ, Yu XL, Mo M, Hu N, Shao ZM, Liu GY. Clinical feasibility and oncological safety of non-radioactive targeted axillary dissection after neoadjuvant chemotherapy in biopsy-proven node-positive breast cancer: a prospective diagnostic and prognostic study. Int J Surg. 2023 Jul 1;109(7):1863-1870. doi: 10.1097/JS9.0000000000000331. PMID 37132193